CLINICAL TRIAL: NCT06671860
Title: Investigation Of The Effects Of Oculomotor Exercises And Hands-On Protocol In Patients With Non-Specific Neck Pain
Brief Title: The Effects Of Oculomotor Exercises And Hands-On Protocol In Non-Specific Neck Pain
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yeditepe University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: Yeditepe U4
Record Dates: First submitted 2024-10-31; First posted 2024-11-04 (Actual); Last update posted 2024-11-04 (Actual); Status verified 2024-10

CONDITIONS: Neck Pain Musculoskeletal
Keywords: neck, non-specific neck pain, exercise, oculomotor exercises, myofascial release
MeSH Terms: conditions — Motor Activity | interventions — Exercise

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Routine Exercise Group The routine exercise program included the following exercises: chin stretchin (Experimental)
  Interventions: Other: Exercise
- Oculomotor Exercise Group The oculomotor exercise program consisted of a series of activities such a (Active Comparator)
  Interventions: Other: Exercise

INTERVENTIONS:
Other: Exercise — Individuals were randomly assigned to the REP (Routine Exercise Program) group and the OHP group. The REP group received the traditional exercise protocol and the OHP group received oculomotor exercises and myofascial release techniques in addition to the traditional exercise. The groups were evaluated before the treatment and at the end of the 6-week treatment sessions. Patient education was given to the patients before both programs. Patient education included information about nonspecific chronic neck pain, symptoms, and complications, as well as assessment methods, parameters, tests, and exercises.
  The first group, the REP group (n=19), received routine exercises, and the second group, the OHP group (n=19), received oculomotor exercises and myofascial relaxation techniques in addition to the routine exercise program. The treatments were applied for six weeks, three sessions per week, under the supervision and guidance of a physiotherapist in the clinic.

SUMMARY:
This study aimed to evaluate the effectiveness of adding oculomotor techniques and hands-on treatments to routine exercise protocols for individuals with non-specific chronic neck pain (NSCNP).

DETAILED DESCRIPTION:
A randomized controlled trial was performed at the orthopedic rehabilitation clinic. Ethical Standards in the 1946 Declaration of Helsinki, as revised in 2013, were followed, and the University Ethics Board approved the study (approval number 147). This research did not receive any specific grant from funding agencies in the public, commercial, or not-for-profit sectors. The study was conducted with individuals aged 18-65 who applied to a private clinic, received a doctor's diagnosis, met the inclusion criteria, and voluntarily agreed to participate in the study.

Participants A total of 38 subjects were calculated as the minimum required sample size determined by power analysis, and 38 subjects aged 18 to 65 years with a diagnosis of nonspecific neck pain who met the inclusion criteria and voluntarily agreed to participate were included in the study. Signed consent forms were obtained from the volunteers who agreed to participate in the study by face-to-face interview.

ELIGIBILITY:
Inclusion Criteria:

* The inclusion criteria included being between ages 18 and 65 old, having been diagnosed with nonspecific neck pain, being able to comply with exercise instructions and understand evaluation questions, and volunteering to participate in the research.

Exclusion Criteria:

History of acute or chronic musculoskeletal pain other than nonspecific neck pain, history of a rheumatological disease, sequestered or extruded disc herniation, having received physical therapy in the last three months, recent history of surgery, infectious and vascular diseases, and cooperation and communication problems presence were excluded.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Estimated)
Dates: Start 2023-06-10 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2024-11-22 (Estimated)

PRIMARY OUTCOMES:
Pain intensity | 6 week
  Pain intensity was measured with a visual analog scale (VAS).

SECONDARY OUTCOMES:
Proprioception | 6 week
  joint position sense (JPS) was assessed using a laser pointer.

CONTACTS AND LOCATIONS:
Locations (1):
- Yeditepe university, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Bier JD, Scholten-Peeters WGM, Staal JB, Pool J, van Tulder MW, Beekman E, Knoop J, Meerhoff G, Verhagen AP. Clinical Practice Guideline for Physical Therapy Assessment and Treatment in Patients With Nonspecific Neck Pain. Phys Ther. 2018 Mar 1;98(3):162-171. doi: 10.1093/ptj/pzx118. PMID 29228289